CLINICAL TRIAL: NCT04017845
Title: Screening for Colorectal Cancer in Average and High Risk Iraqi Population: A Pilot Study
Brief Title: Screening for Colorectal Cancer in Average and High Risk Population
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lewai Sharki Abdulaziz, MSc PhD (Other)
Collaborators: Research & Development Directorate, Ministry of Higher Education, Iraq (Unknown); Al-Kindy College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Lewai Sharki Abdulaziz, MSc PhD, Assistant Professor, Al-Kindy College of Medicine
Organization: Al-Kindy College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 3Al-KindyCM
Record Dates: First submitted 2019-07-01; First posted 2019-07-12 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer; Adenomatous Polyp of Colon
Keywords: Colorectal cancer; Screening; Fecal Immunochemical Test
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tribenoside; Lidocaine; Suppositories; tribenoside (combination); Diltiazem; Calcium Channel Blockers; Nitrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Household-Open Invitation (HOI) (Active Comparator): Precolonoscopy cleansing regimen and referral to conventional colonoscopy is based on Positive FIT (level ≥75ng/ml) in any of the two collected samples. Histopathological examinations of screen-detected lesions are reported and lesion with the worst prognosis is indicated as the final colonoscopic outcome used for evaluation purposes. Screenees with intermediate and high risk polyp were referred to a follow-up surveillance programme.Treatments were initiated with Diltiazem hydrochloride 2%/Nitroglycerin rectal ointment for anal fissure, and tribenoside 400 mg + lidocaine 40 mg suppositories for hemorrhoids. Positive FIT results in participants who were identified with no adenomas, advance adenomas, or adenocarcinomas are considered False-positive FIT (FP-FIT) results.
  Interventions: Diagnostic Test: FIT; Procedure: Precolonoscopy cleansing regimen; Procedure: Conventional Colonoscopy; Diagnostic Test: Histopathological examinations of screen-detected lesions; Drug: Tribenoside 400 mg + lidocaine 40 mg suppositories; Drug: Diltiazem hydrochloride 2%/Nitroglycerin rectal ointment
- Recommendation By Physician (RBP) (Active Comparator): Precolonoscopy cleansing regimen and referral to conventional colonoscopy is based on Positive FIT (level ≥75ng/ml) in any of the two collected samples. Histopathological examinations of screen-detected lesions are reported and lesion with the worst prognosis is indicated as the final colonoscopic outcome used for evaluation purposes. Screenees with intermediate and high risk polyp were referred to a follow-up surveillance programme.Treatments were initiated with Diltiazem hydrochloride 2%/Nitroglycerin rectal ointment for anal fissure, and tribenoside 400 mg + lidocaine 40 mg suppositories for hemorrhoids. Positive FIT results in participants who were identified with no adenomas, advance adenomas, or adenocarcinomas are considered False-positive FIT (FP-FIT) results.
  Interventions: Diagnostic Test: FIT; Procedure: Precolonoscopy cleansing regimen; Procedure: Conventional Colonoscopy; Diagnostic Test: Histopathological examinations of screen-detected lesions; Drug: Tribenoside 400 mg + lidocaine 40 mg suppositories; Drug: Diltiazem hydrochloride 2%/Nitroglycerin rectal ointment

INTERVENTIONS:
Diagnostic Test: FIT — Screenees were supplied with two fecal collection devices and asked to collect two specimens from two consecutive Different Bowel Movement Samples (DBMS) or, in case of infrequent bowel movements, from the Same Bowel Movement Sample (SBMS).Instruction stressed that after collection the device must be stored in refrigerator and transported in an iced pack within no more than 48h from sampling. After checking for sampling appropriateness, the received samples were analyzed by the FOB Gold/SENTiFOB method (Sentinel Diagnostics SpA, Milan, Italy), according to the previously validated procedural platform
  Other Names: Fecal Immunochemical Test (FIT); Fecal occult blood tests (FOBT); FOB Gold/SENTiFOB (Sentinel Diagnostics SpA, Milan, Italy)
Procedure: Precolonoscopy cleansing regimen — Laxative stimulant two days prior to the cleansing regimen involves the intake of one 10 mg tablet of bisacodyl (Dulcolax, Sanofi,UK) at 18:00 for two consecutive nights.The evening before colonoscopy cleansing started with 2 doses (at 16:00 and 20:00) of one sachet Sodium picosulphate preparations (PICOPREP, Ferring Pharmaceutical Co., Ltd., Zhongshan, China), dissolved in150 mL of cold water, followed with five 240 mL portions of clear liquids within 3 h. The third dose is taken in the morning about 5 h prior to colonoscopy, followed with at least three 240 mL portions of clear liquids no later than 2 h before colonoscopy.
  Other Names: PICOPREP- Adjuvant Bisacodyl Regimen
Procedure: Conventional Colonoscopy — With the colonoscopists completely blinded regarding the FIT results, conventional colonoscopy examinations were conducted in the Endoscopy Unit of Al-Kindy Polyclinic. According to the five levels of competency proposed by the European guidelines, this unit is assigned as level 2, with the possibility of removing polypoid and sessile lesions <25 mm, providing there is good access. For flat lesions, larger sessile and polypoid lesions, and smaller lesions with more difficult access, the lesions were documented appropriately with the patients referred to higher competent units in order to be safely and expertly removed.
  Other Names: Optical Colonoscopy
Diagnostic Test: Histopathological examinations of screen-detected lesions — Adenomas were classified according to the modified revised Vienna classification for the European Guidelines. Advanced adenoma was defined as the presence of one of the following features: >10 mm diameter, tubulovillous or villous structure, and high-grade neoplasia. Polypoid adenocarcinomas were reported according to the TNM classification, while colorectal cancer associated with flat and/or depressed lesions were reported as non-polypoid lesions, and further classified by the Paris classification. Pathologic results of hyperplastic polyps, sessile serrated lesions or post inflammatory polyps were considered normal findings.
  Other Names: Histological examinations of Lesion Biopsies and Resections
Drug: Tribenoside 400 mg + lidocaine 40 mg suppositories — Treatment of hemorrhoids was initiated with tribenoside 400 mg + lidocaine 40 mg suppositories, once daily for up to 2 weeks.
  Other Names: PROCTO-GLYVENOL
Drug: Diltiazem hydrochloride 2%/Nitroglycerin rectal ointment — Treatment of anal fissure was initiated with Diltiazem hydrochloride 2%/Nitroglycerin rectal ointment applied every 12 hours, for up to six weeks.
  Other Names: Topical calcium channel blockers/nitrates

SUMMARY:
The existing evidence from epidemiological studies and randomized controlled trials has consistently assures the cost effectiveness and the influential role of screening in reducing incidence rates and deaths caused by Colorectal Cancer (CRC). Population based organized screening programmes, which should be considered an obligation that is not to be postponed, require valuable information that can be reliably extrapolated from well-designed pilot study conducted prior to programme implementation.

The main objectives of the current pilot CRC screening project, named after "Al-Kindy College of Medicine", was to evaluate and explore the specific aspects of the intended population-based organized CRC screening programme, including: barriers affecting adherence to the programme, performance indicators of the proposed screening programme, the target population in which CRC screening is a legitimate healthcare priority, quality assurance of screening tests and colonoscopy services, and to propose an algorithm that will provide a clinically and logistically acceptable positivity rate.

DETAILED DESCRIPTION:
Screening Type and Setting :

"Al-Kindy College Colorectal Cancer Screening Project", is proposed as an FIT-based colorectal cancer screening, with colonoscopy being used as the second stage investigation in those with a positive FIT result. This screening project was set as a 24 months pilot study, to be started in April 2015 and extended to May 2017. All the investigations and evaluation measures involved were performed in the scientific research laboratory and endoscopy unit of Al Kindy polyclinic at Al Kindy College of Medicine, University of Baghdad. Baghdad, Iraq.

Study Protocol:

Target Individuals and Eligibility:

The target individuals of the present study are residents of Baghdad city being ≥45 years of age with stop age of 80 years. target individual with fulfill devoid of exclusion criteria is identified as eligible.

Invitation of Eligible Individuals:

Due to the lack of a population register, invitation for the proposed screening programme was based on two approaches, namely, household open invitation (HOI), and recommendation by physician (RBP).

1. Household-Open Invitation (HOI): A survey sheet, which all together serves as an invitation letter, was assembled competently. The first part of the sheet, in Arabic language, included introductory information about CRC incidence and risk factors, CRC screening benefits and meaning of test results, along a briefly description for the potential diagnostic tests and treatment options. The second part aimed to document information about the invited families, including demographic data, the number of target individuals and their eligibility, as well as the prevalence of CRC risk factors including: body mass index (BMI), smoking and alcohol intake, type2 diabetes mellitus (T2DM) and family history of CRC. Total of 1000 survey sheets were delivered by 10 teams, each team consist of 10 well-trained 4th stage students of Al Kindy College of Medicine, as part of their epidemiology training course. The dissemination was planned, in an order of 100 families per week, with as possible equity to ensure the coverage of all municipalities of Baghdad city. Students were requested to return the day next to delivery, to check for the eligibility of target individuals and participation consent.
2. Recommendation By Physician (RBP): A random survey of 1000 outpatients, attending Endocrine Disease Treatment Center, Baghdad, Iraq, was arranged with the aim of encouraging patients who fulfil the criteria for eligibility to participate in the screening programme. Referral forma including participation consent was issued, as an act on acceptance, and the issued referral forma were documented to measure patients' compliance.

Enrollment of Participants in the Proposed Screening Programme:

Screenees' basic information and progressive examination outcomes were documented through a comprehensive "Audit and Tracking Sheet", divided into the following four major disciplines:

1. Characteristics and Risk Stratification:

   To evaluate the impact of risk stratification on screenee's behavior and on the effectiveness of the screening project, participants were divided into three risk groups based on survey and medical record data: high-risk (history of polyps, and/or personal/family history of CRC, increased-risk (diabetes, obesity, and/or former or current smoking status), and average-risk (45 or older with no other risk factor).
2. FIT and Colonoscopy Tracking Screening Schedule:

   After checking for sampling appropriateness, the received samples were analyzed by the FOB Gold/SENTiFOB method (Sentinel Diagnostics SpA, Milan, Italy), according to the previously validated procedural platform.

   In case of first FIT incompletion, the cause is identified and the screenees were encouraged for re-enrollment. Timely referral to colonoscopy was based on FIT level ≥75ng/ml in any of the two collected samples. Negative FIT-tested individuals with high risk stratification were also encouraged to be enrolled. On approval, after a brief elucidation for the pros and cons, screenees were scheduled for conventional colonoscopy.

   Considering the reported improved patient tolerance of sodium picosulphate preparations (PICOPREP, Ferring Pharmaceutical Co., Ltd., Zhongshan, China), this cleansing agent was preferentially prescribed.Detailed oral and written instructions on how to perform the bowel cleansing regimen was provided, with an excellent opportunity to answer any questions the screenee may have, to ensure that the process was appropriately understood.

   With the colonoscopists completely blinded regarding the FIT results, conventional colonoscopy examinations were conducted in the Endoscopy Unit of Al-Kindy Polyclinic. For non-compliance, the cause of cancelled appointment was identified, and screenees were reinvigorated for a rescheduled appointment. For attendants, on the other hands, the final examination report must verify the completeness of colonoscopy; otherwise, the report should point to the cause of incompleteness. The report should also document the number, size, type and anatomical location of any screen-detected lesions.
3. Histological Report of Lesion Biopsies and Resections:

   Histopathological examinations of screen-detected lesions were performed by skilled pathologists in gastrointestinal disease with specific emphasis on colorectal cancer, along a good expertise in the preparation and interpretation of biopsies and endoscopic polypectomy specimens.

   Classification of adenomas included grading of neoplasia was accomplished according to the revised Vienna classification that has been modified for the European Guidelines to obtain a two- tiered system of low-grade and high-grade neoplasia.. Furthermore, and whenever applicable, the correlation between histological diagnosis of biopsy and resection specimens were included in the final examination reports.

   If more than one lesion is found, lesion with the worst prognosis is indicated as the final colonoscopic outcome and will be used for evaluation purposes. Based on the number and characteristics of adenomas detected at baseline colonoscopy, screenees were stratified into low, intermediate, and high risk polyp for the development of colorectal cancer. Screenees with intermediate and high risk were referred to a follow-up surveillance programme. Positive FIT results in participants who were identified with no adenomas, advance adenomas, or adenocarcinomas on subsequent colonoscopies are considered False-positive fecal immunochemical tests (FP-FIT) results.
4. Quality Assurance of Screening Programme:To ensure a potential benefit of colorectal cancer screening, quality assurance of the programme was assessed at every step in the process, including the FIT sampling regimen, precolonoscopy cleansing regimen, bowel preparation quality using the Ottawa bowel preparation scale (OBPS), as well as colonoscopy quality with special emphasis on colonic mucosa inspection and the safety and tolerance of colonoscopy.

Data Processing and Statistical Analysis:

All Data analysis was processed by the statistical package SPSS version 21.0 (SPSS, Inc.). Descriptive and categorical variables were presented as frequencies and percentages, and Fischer's exact test was performed to inspect any association between these variables. Indicators of screening performance for FIT (including participation rate, and positivity rate) and colonoscopy (including compliance rate, completion rate, lesions detection rate, adenoma detection rate, advanced adenoma detection rate, and cancer detection rate), in addition to the positive predictive value (PPV) for detection of lesions, adenoma, advanced adenoma, and cancer, were all calculated according to the European guidelines for quality assurance in colorectal cancer screening and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* residents of Baghdad city
* being ≥45 years of age with stop age of 80 years.

Exclusion Criteria:

* history of inflammatory bowel disease (IBD).
* colonoscopy (CS)/flexible sigmoidoscopy (FS)/ double contrast barium enema (DCBE) performed within the last year.
* persistent altered bowel habits.
* chronic abdominal pain.
* visible bleeding per rectum.
* long term use of anticoagulant.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
prevalence of causes accounting for population disagreement to participate in screening. programme. | Documented on one occasion, during invitation interview as an act on disagreement to participate in the screening programme.
  Eligible screenees who do not have the willingness to participate were asked to identify their disagreement cause(s) from the list included in the invitation letter and reported as:
  1. I don't have the will or time to be enrolled.
  2. My residence is far off the program center.
  3. I am afraid the program will unveil the presence of the disease.
  4. I cannot accept and tolerate the tests included in the program.
  5. I am not fully persuaded about the program achievability.
  6. Infeasibility of freely provided medical services.
Prevalence of CRC risk factors and risk stratification in target population. | Documented on one occasion, during invitation interview, as an act on agreement to participate in the screening programme.
  individuals of the target population were divided into three risk groups based on survey and medical record data: high-risk (history of polyps, and/or personal/family history of CRC, increased-risk (diabetes, obesity, and/or former or current smoking status), and average-risk (45 or older with no other risk factor).
Performance Indicators of Fecal Immunochemical Test (FIT) | Documented on one occasion, immediately after completion of FIT testing.
  the performance of Fecal Immunochemical Test (FIT) during the screening process was assessed in terms of participation rate,completion rate and positivity rate.
Performance Indicators of Colonoscopic Examination | Documented on one occasion, immediately after completion of colonoscopy examination.
  the performance of follow up colonoscopy during the screening process was assessed in terms of referral rate, compliance rate, completion rate and lesion detection rate.

OTHER OUTCOMES:
Quality assurance of Fecal Immunochemical Test (FIT): short questionnaire | Documented on one occasion, immediately after completion of FIT testing.
  Quality assurance of the Fecal Immunochemical Test (FIT) was assessed by a short questionnaire related to the sampling and testing process including:
  1. the ease of use of FOB Gold Tube NG fecal collection device.
  2. the suitability of the post-sampling storage and transportation processes.
  3. the number of unacceptable specimens due to sample error or delay.
  4. the number of received samples appropriately analyzed within the time specified in study protocol.
Quality assurance of precolonoscopy cleansing regimen: Ottawa Bowel Preparation Scale (OBPS) | Documented on one occasion, immediately after completion of colonoscopy examination.
  The precolonoscopy cleansing regimen was assessed according to the quality of bowel preparation for colonoscopies using the total Ottawa Bowel Preparation Scale (OBPS).The scale individually assesses three parts of the colon: (1) the right colon, (2) the middle colon and (3) the rectosigmoid colon. Subscores of 0 to 4 were used for each section of the colon, along with a fourth separate subscore of 0 to 2 for overall fluid .These four individual subscores are added, and the total score of between 0 and 14 provides an assessment of bowel preparation quality, which is judged as:
  1. An excellent bowel preparation has a total score of 0 to 1.
  2. A good bowel preparation has a score of 2 to 4.
  3. A fair bowel preparation has a score of 5 to 7.
  4. A poor bowel preparation has a score of 8 to 10.
  5. An inadequate bowel preparation has a score of 11 to 14.
Safety and tolerance of precolonoscopy cleansing regimen: short questionnaire | Documented on one occasion, immediately after completion of colonoscopy examination.
  Safety and tolerance of precolonoscopy cleansing regimen was assessed by a short questionnaire including:
  1. frequency and severity of associated symptoms.( nausea, vomiting, chest pain, abdominal cramps and abdominal distension).
  2. frequency of related complications ( electrolytes imbalance, dehydration, brief loss of consciousness, convulsions, syncope and ischemic colitis).
  3. ability to complete bowel preparation.
  4. willingness to repeat the same bowel preparation.
Quality assurance of colonoscopic examination: rates of ceacal intubation and the lesions detection rate | Documented on one occasion, immediately after completion of colonoscopy examination.
  The quality of colonoscopic examination was assessed according to the rates of ceacal intubation and the lesions detection rate.
safety and tolerance of colonoscopy. | Documented on one occasion, immediately after completion of colonoscopy examination.
  Safety and tolerance of colonoscopy examination was assessed by a short questionnaire including:
  1. frequency and severity of associated discomfort and or abdominal pain.
  2. frequency of related complications ( cardio-respiratory event, perforation, bleeding and infection).
  3. ability to complete colonoscopy examination.
  4. willingness to repeat the same colonoscopy examination.

CONTACTS AND LOCATIONS:
Overall Officials: Lewai S Abdulaziz, MSc PhD, Study Chair — Al-Kindy college of Medicine, University of Baghdad; Faris A Khazaal, FRCP, Principal Investigator — Al-Kindy college of Medicine, University of Baghdad; Riyadh M Hasan, CABS, Principal Investigator — Al-Kindy college of Medicine, University of Baghdad; Mohammed A Al-Kurtas, FICMS.Path, Principal Investigator — Al-Kindy college of Medicine, University of Baghdad
Locations (1):
- Lewai S Abdulaziz, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No